CLINICAL TRIAL: NCT05212662
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Study to Assess the Safety, Tolerability, Pharmacodynamics (PD) and Efficacy of TTI-0102 for the Treatment of Patients With Mild to Moderate COVID-19
Brief Title: Study of Cysteamine-pantetheine Disulfide (TTI-0102) in Mild to Moderate COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor is not pursuing the COVID-19 indication at this time.
Sponsor: Thiogenesis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTI-CV-001
Record Dates: First submitted 2022-01-26; First posted 2022-01-28 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: COVID-19; COVID-19 Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19 | interventions — cysteamine-pantetheine disulfide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TTI-0102 (Experimental): Cysteamine-pantetheine disulfide (TTI-0102) is supplied in a vial as a powder to be dissolved in water and administered orally.
  Interventions: Drug: TTI-0102
- Placebo (Placebo Comparator): Placebo is supplied in a vial as a powder to be dissolved in water and administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TTI-0102 — The study treatment is a precursor to cysteamine, TTI-0102 (cysteamine-pantetheine disulfide). Each molecule of TTI-0102, after reduction and metabolism in the digestive tract, allows the absorption of 2 molecules of cysteamine and one molecule of pantothenic acid (Vit B5). Each dose of TTI-0102 comes in a vial as a powder to dissolve in water and absorb orally. Each vial contains 5.5g of TTI-0102, corresponding to the equivalent of 2.4g of cysteamine base. This single dose is less than the maximum daily dose authorized with other formulations of cysteamine (Cystagon or Procysbi, 1.95 g/m2/day) for patients over 1.25 m2 or 40 kg (88 lbs).
  This dose of 5.5 g is justified by the need to maintain a thiol/disulfide ratio in favor of cysteamine over 24 h. It has been tested in healthy volunteers and has no side effects due to the specific pharmacokinetics of cysteamine after administration of TTI-0102.
  Other Names: cysteamine-pantetheine disulfide
  Arms: TTI-0102
Drug: Placebo — Placebo comparator supplied in vials identical to the active intervention, TTI-0102
  Arms: Placebo

SUMMARY:
This is multi-center, randomized, double-blind, placebo-controlled study to assess the safety, tolerability, pharmacodynamics (PD) and efficacy of TTI-0102 for the treatment of patients with mild to moderate COVID-19. This is a phase 2 study of cysteamine-pantetheine disulfide (TTI-0102), an antiviral, anti-infectious, antioxidant and anti-CRS (cytokine release syndrome) investigational drug. Subjects will be randomized 2:1 to receive TTI-0102 or placebo daily for up to 14 days. Up to 5 centers in the US and Canada will conduct this study. 60 patients will be enrolled.

DETAILED DESCRIPTION:
All patients with confirmed COVID-19 will be managed within an outpatient continuum of care management program that includes self-assessment tools; initial telephone triage; coordinated outreach and management approach based upon individual patient risk, severity of symptoms, and time course of disease; clinician telehealth (telephone call or video platform-based) visits (initial evaluation and follow-up visits); COVID-19 testing; a separate outpatient respiratory clinic or dedicated space within an ambulatory clinic appropriated for the care of patients with COVID-19 and other respiratory problems; strategies to reduce the risk of exposure to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) by staff and other patients will be employed.

Screening Period - Remote Patients will undergo screening to determine study eligibility, for a period of not more than 7 days. It is not required that patients come to study investigator clinic for screening assessments, but SARS-CoV-2 PCR test results, medical history and vital signs used to verify study eligibility must be collected from the non-investigator facility that performed them, reviewed prior to Day 1, placed in the subjects' source documentation and transcribed to the CRF. The Ethics Committee or Institutional Review Board must approve the informed consent template and the remote consent process and documentation to be utilized for the trial.

Treatment Period (Days 1-14)

* Day 1 Clinic Visit: Eligible subjects will be enrolled into the study, i.e. randomization will take place, they will receive their first dose of study drug (TTI-0102 or placebo) in clinic, and they will be dispensed enough to continue treatment at home for up to 14 days. Baseline assessments will be performed according to Appendix 22.1 Schedule of Assessments.
* Day 8 - Remote Visit: Subjects will be contacted to assess their tolerance to study drug. Subjects unable to tolerate the 5.5 gram daily dose (QD) will be instructed to split the dose into two 2.75 gram half-doses taken in the morning and the evening (BID).
* Day 14 - Clinic Visit: Subjects will return to clinic for end-of-treatment assessments specified in Appendix 22.1 Schedule of Assessments.

Subjects will continue daily study drug treatment as outpatients, under home quarantine as per local Public Health guidelines. Subjects will also receive continued standard of care therapy per study site written policies or guidelines. Study drug treatmetn should continue for 14 days, or earlier as medically appropriate (e.g., deterioration of clinical status and alternative therapy required). If the patient requires hospitalization during the study period, study drug treatment will be discontinued.

The following safety assessments will be performed at timepoints specified in the Appendix 22.1 Schedule of Assessments. In addition to unsolicited, spontaneous adverse events which are reported or observed, patients will be interviewed for additional cysteamine-associated adverse events using a protocol-specific checklist [Appendix 22.8]. Subjects will also be asked to complete the Gastrointestinal Symptom Rating Scale (GSRS) [Appendix 22.7] and a COVID-19 symptoms questionnaire [Appendix 22.6].

If a patient is required to show up in an outpatient clinic, physical examinations, electrocardiograms (ECGs), vital signs, and clinical laboratory evaluations (chemistry, hematology, urinalysis) will be performed. A standardized toxicity grading scale will be used to grade the severity of adverse events, National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) [Appendix 22.9].

Study Termination: Day 28 or upon Early Withdrawal - Remote Visit A remote (telephone or video) Study Termination Visit will take place on Day 28 for patients who completed treatment or, for patients who withdraw early, 2 weeks (14 days) after the last study drug dose.

Follow-up Period - Remote Visits Follow-up telephone contact #1 will be performed on Day 42 or 28 days/4 weeks after last study drug dose. Follow-up telephone contact #2 will take place on Day 70, or 56 days/7 weeks after last study drug dose.

ELIGIBILITY:
Inclusion Criteria:

1. Is between 18 and 80 years of age.
2. Is within 72 hours from onset of symptoms consistent with COVID-19 at time of study screening.
3. Has at least 2 of the following: fever (oral temperature ≥38°C), cough, shortness of breath, chest x-ray changes consistent with COVID-19 at time of screening.
4. Has a laboratory-confirmed SARS-CoV-2 infection as determined by FDA-approved rapid diagnostic (e.g., PCR) assay.
5. Has a score of ≤ 2 on the 8-category National Institute of Allergy and Infectious Diseases (NIAID) ordinal rating scale at time of screening. [Protocol Appendix 22.2]
6. Agrees to the collection of blood and urine samples, nasopharyngeal (NP) swabs, and non-invasive oxygen monitoring (via pulse oximeter) as required by study protocol.
7. Patient or their legally authorized representative is willing and able to provide written informed consent prior to performing study procedures.
8. Understands and agrees to comply with planned study procedures.
9. Women of childbearing potential must agree to either abstinence or use of at least one primary form of contraception not including hormonal contraception from the time of screening through Day 29 following randomization. All subjects of childbearing potential, including males with partners of childbearing potential, must use highly effective methods of birth control defined as those, alone or in combination, that result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly [Protocol Appendix 22.3]. Abstinence is NOT an acceptable method of contraception UNLESS it is the subject's normal practice

Exclusion Criteria:

1. Is currently hospitalized.
2. Prior history of, or considered to be at risk for, agranulocytosis, nephropathy, liver disease or interstitial pneumonia.
3. Current or historic positive human immunodeficiency virus (HIV) test.
4. Presence of organ transplant.
5. Receipt of cancer chemotherapy or immunomodulatory drugs including but not limited to biologics such as anti-CD20, anti-TNF, anti-IL6; alkylating agents (e.g., cyclophosphamide), antimetabolites (e.g., azathioprine), or chronic corticosteroid use equivalent to prednisone >10 gm/day, during the 2 months prior to screening.
6. Confirmed positive for influenza at screening.
7. Confirmed positive for respiratory syncytial virus (RSV) at screening.
8. Pregnant or breastfeeding.
9. Current use of, or known allergy to cysteamine, bucillamine or penicillamine (e.g., for Wilson's disease, rheumatoid arthritis).
10. Current participation in any other clinical trial of an experimental treatment for any indication including COVID-19.
11. Receipt of any experimental treatment for COVID-19 (herbal, homeopathic, over the counter, off-label, compassionate use, or clinical trial related) within the 30 days prior to screening.
12. Receipt of any medication for treatment or prevention of COVID-19 being used pursuant to an Emergency Use Authorization (e.g., vaccine) prior to or during study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09-27 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint | 28 days
  Frequency of hospitalization or death

SECONDARY OUTCOMES:
Secondary: Safety | 28 days
  Frequency of adverse events
Secondary: Efficacy | 28 days
  Change of COVID-19 symptoms (self-assessment) score from Baseline, as measured at Day 14 and Day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Patrice P Rioux, MD, PhD, Study Director — Sponsor: Thiogenesis Therapeutics, Inc.

IPD SHARING:
Plan to Share IPD: No